CLINICAL TRIAL: NCT04044404
Title: Application of Ultrasound Integrated Precision Diagnosis Technology in Prevention of Kidney Disease and Its Progress
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: RJ2018049; 2019-52-K33 (Other: China-Japan Friendship Hospital)
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Diagnostic Imaging; Diagnosis; Kidney Disease
Keywords: Ultrasound Elastography; Ultrasound Integrated Precision Diagnosis Technology; Acute on Chronic Kidney Disease; Kidney transplantation; kidney fibrosis
MeSH Terms: conditions — Disease; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A on C group: Acute on Chronic Kidney Disease patients
  Interventions: Diagnostic Test: Ultrasound Integrated Precision Diagnosis Technology(ultrasound elastography)
- functional delayed graft function group: patients with functional delayed graft function(fDGF) after kidney transplantation
  Interventions: Diagnostic Test: Ultrasound Integrated Precision Diagnosis Technology(ultrasound elastography)
- Normal: without functional kidney injury
  Interventions: Diagnostic Test: Ultrasound Integrated Precision Diagnosis Technology(ultrasound elastography)

INTERVENTIONS:
Diagnostic Test: Ultrasound Integrated Precision Diagnosis Technology(ultrasound elastography) — Compare the ultrasound Integrated Precision Diagnosis Technology(ultrasound elastography) with the diagnostic gold standard of kidney disease---kidney biopsy

SUMMARY:
In this study, a prospective, randomized and controlled clinical study would be carried out to establish Ultrasound Integrated Precision Diagnosis Technology with elastography as the core technology to evaluate renal injury and repair comprehensively and accurately, and to improve the clinical diagnosis chance of renal injury (or renal fibrosis).

Combined with the dynamic changes of biomarkers (inflammatory factors, cytokines secreted by immune cells, etc.) after kidney injury, the research on the prognosis of kidney disease with ultrasound elastography technology as the core would be explored, which aims to provide a scientific basis for the application of Ultrasound Integrated Precision Diagnosis Technology.

ELIGIBILITY:
Inclusion criteria

1. for A on C group 1.18-70 years old; gender is not limited; 2. Patients who can cooperate with breath-holding, breath-holding and breath-exhaling movements, and communicate without obstacles.

   3.The informed consent has been signed; 4.Abnormal renal pathology or glomerular filtration rate(GFR) (15 <GFR<90 ml/min.1.73 m2) or proteinuria > 1 g/24 h due to any cause.
2. for kidney transplantation

   1. 18-70 years old; gender is not limited;
   2. It can cooperate with breath-holding, breath-holding and breath-exhaling movements, and communicate without obstacles.
   3. The informed consent has been signed;
   4. Kidney transplant recipients in our hospital from May 2019 to November 2019

Exclusion criteria

1. for A on C group

   1. Can't cooperate, can't lie down for at least 10 minutes, unconsciousness, severe hypoxia, restlessness need to rescue patients.
   2. Patients with pregnancy or cancer;
   3. There are other serious diseases that the researchers do not think it is suitable to participate in this experiment.
   4. Absolute contraindications of renal puncture, ① Obvious bleeding tendency; ②Severe hypertension (systolic pressure greater than 180 mm Hg or diastolic pressure greater than 115 mm Hg); ③Psychiatric patients or non-cooperating operators and isolated kidney (small kidney) Or relative contraindications of renal puncture: ① Active pyelonephritis, renal tuberculosis, hydronephrosis or pyonephrosis, ②renal abscess or perirenal abscess. ③Renal tumors or renal aneurysms. ④Polycystic kidney or renal cyst. ⑤Kidney position is too high (deep inhalation of the lower pole of the kidney is not below the twelve ribs) or migratory kidney. ⑥Obesity, severe ascites.

      b）for kidney transplantation

   <!-- -->

   1. Can't cooperate, can't lie down for at least 10 minutes, unconsciousness, severe hypoxia, restlessness need to rescue patients.
   2. Patients with pregnancy or cancer;
   3. There are other serious diseases that the researchers do not think it is suitable to participate in this experiment.
   4. Absolute contraindications of renal puncture, ① Obvious bleeding tendency; ②Severe hypertension (systolic pressure greater than 180 mm Hg or diastolic pressure greater than 115 mm Hg); ③Psychiatric patients or non-cooperating operators and isolated kidney (small kidney) Or relative contraindications of renal puncture: ① Active pyelonephritis, renal tuberculosis, hydronephrosis or pyonephrosis, ②renal abscess or perirenal abscess. ③Renal tumors or renal aneurysms. ④Polycystic kidney or renal cyst. ⑤Kidney position is too high (deep inhalation of the lower pole of the kidney is not below the twelve ribs) or migratory kidney. ⑥Obesity, severe ascites.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For A on C group:18-70 years old patient who can cooperate with breath-holding, breath-holding and breath-exhaling movements, and communicate without obstacles, signed informed consent and with abnormal renal pathology or glomerular filtration rate(GFR) (15 <GFR<90 ml/min.1.73 m2) or proteinuria > 1 g/24 h due to any cause.
  For fDGF in kidney transplantation patient :18-65 years old patient who can cooperate with breath-holding, breath-holding and breath-exhaling movements, and communicate without obstacles, signed informed consent and received Kidney transplant recipients in our hospital from May 2019 to November 2019.
Sampling Method: Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-05-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with creatinine increasing by more than 50% | 1st month-12 month
  Number of patients with creatinine increasing by more than 50% of baseline.
Number of patients with initiation of continuous renal replacement therapy | 1st month-12 month
  for non-transplantation patient
Rate of death | 1st month-12 month
  for all patients

SECONDARY OUTCOMES:
Number of patients with cardiovascular events | 1st month-12 month
  (acute myocardial infarction, unstable angina pectoris, heart failure requiring hospitalization or death from cardiovascular diseases);
Number of patients with cerebrovascular events | 1st month-12 month
  (cerebral hemorrhage, subarachnoid hemorrhage, ischemic stroke, transient ischemic attack or death from cerebrovascular diseases);
Number of patients with new serious infections requiring hospitalization | 1st month-12 month
  for all kidney injury

OTHER OUTCOMES:
Number of patients with recovery of creatinine within 7 days less than 70%. | 1st month-12 month
  for renal transplantation patient
Number of patients with allograft loss | 1st month-12 month
  for renal transplantation patient

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of nephrology , Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - China-Japan Friendship Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No